CLINICAL TRIAL: NCT00143702
Title: Randomized, Open-Label Study of Continued Stavudine Versus Abacavir Substitution With or Without Riboflavin and Thiamine Supplementation in HIV-Infected Patients Who Have Elevated Venous Lactic Acid While on Stavudine-Based Therapy (DAVE)
Brief Title: D4T or Abacavir Plus Vitamin Enhancement in HIV-Infected Patients (DAVE)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: GlaxoSmithKline (Industry); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Dr. Julio Montaner, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P00-0159; CTN 169
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2005-09

CONDITIONS: Acidosis, Lactic
Keywords: Elevated Lactic Acid
MeSH Terms: conditions — Acidosis, Lactic | interventions — Stavudine; abacavir; Riboflavin; Thiamine; Dietary Supplements

INTERVENTIONS:
Drug: d4T — See Detailed Description.
Drug: Abacavir — See Detailed Description.
Drug: Riboflavin and Thiamine (Supplementation) — See Detailed Description.

SUMMARY:
The purpose of this study is to determine the best way to treat people on d4T (stavudine) with high levels of lactic acid. Switching from d4T to abacavir will be assessed. Adding riboflavin and thiamine will also be assessed.

Participants will be randomly assigned to one of four groups:

* Group 1 participants will continue to take d4T as part of their antiretroviral (ARV) regimen, and will be given the vitamin supplements
* Group 2 will continue to take d4T without vitamin supplements
* Group 3 will switch from d4T to abacavir and receive the vitamins
* Group 4 will switch from d4T to abacavir without vitamin supplements.

The study plans to involve eighty participants from Canada and Argentina for a treatment period of 16 weeks and a follow-up visit at week 24.

ELIGIBILITY:
Inclusion Criteria:

* Be HIV-positive
* Be 18 years of age or older
* Have a viral load equal to or below 50 copies/mL
* Have been on a d4T-containing multiple drug regimen (at least three agents in total) for at least six months
* Have been on a stable ARV regimen for the three months prior to enrollment
* Have a venous lactic acid measurement above 2.1 mmol/L within the three months prior to enrollment and two consecutive measurements above 2.1 but lower than 6.0 within a two-week period of screening
* Be willing to discontinue L-carnitine and/or coenzyme Q10
* Be willing and able to provide informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Venous lactic acid equal to or above 6.0 mmol/L
* Previous exposure to abacavir
* Virologic rebound while on a previous regimen consisting of dual or triple nucleoside reverse transcriptase inhibitors (NRTIs)
* Use of hydroxyurea within the three months prior to enrollment
* Use of metformin
* Any acute cardiopulmonary illness or infection
* New AIDS-defining illness diagnosed within four weeks of enrollment
* Riboflavin or thiamine supplementation above 20 mg/day within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2001-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients per arm with random venous lactic acid (RVLA) below or equal to 2.1 mmol/L* at 16 weeks. (* Confirmed by a second determination 7-14 days later.) | 16 weeks

SECONDARY OUTCOMES:
Rate of decline of RVLA levels
Absolute level of change of RVLA levels using baseline values as a covariant
Proportion of patients improving/normalizing exercise testing mitochondrial dysfunction pattern
Time to event: time to normalize venous lactic acid
Time to event: premature therapy discontinuation, viral load rebound, and progression to a new AIDS defining illness or death
Proportion of patients with at least three consecutive HIV-1 RNA determinations equal to or below 50 copies/mL during the 16 week follow-up period on an intention to treat basis | 16 weeks
Change in absolute CD4 from baseline
Absolute CD4/CD8 counts
Incidence of grade III and greater adverse drug effects
Metabolic laboratory assessments (anion gap, lipid and hepatic profile, and hematology)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Montaner, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Positive Care Clinic, Toronto, Ontario